CLINICAL TRIAL: NCT02195063
Title: Survey of Patients Who Have Been Prescribed a Topical Compound for Pain Management, Wound Care or Scar Care or to Patients Who Have Been Requested to do a Urinary Drug Test (UDT) by Their Provider.
Brief Title: Survey Study for Pain Management, Wound Care, Scar Care or UDT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rahm Foundation (Other)
Collaborators: Datum Research, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: RAHM 1001
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Scars; Wounds; Urinary Drug Testing
Keywords: Pain management; Scar care; Wound care; UDT; Urinary drug testing
MeSH Terms: conditions — Pain; Cicatrix; Wounds and Injuries; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pain management: patients undergoing transdermal treatment for pain
- Scar care: patients undergoing transdermal treatment for scars
- Wound care: patients undergoing transdermal treatment for wounds
- UDT: patients receiving urinary drug tests

SUMMARY:
This is a survey study that will be given to patients who have been prescribed a topical compound for pain management, wound care or scar care or to patients who have been requested to do a urinary drug test (UDT) by their provider.

The initial survey for pain management, wound care, scar care or UDT will be given to the patient by their providers during their office visit.

DETAILED DESCRIPTION:
We have designed a survey study that will be given to patients who have been prescribed a topical compound for pain management, wound care or scar care or to patients who have been requested to do a urinary drug test (UDT) by their provider.

The initial survey for pain management, wound care, scar care or UDT will be given to the patient by their providers during their office visit.

Follow-up surveys will be given at 30, 60, and 90 days. These surveys will be collected by e-mail or follow-up calls from Datum Research, LLC, contract research organization.

Data collection for this study will be derived through the 4 patient surveys (initial, 30 day, 60 day, and 90 day) and the prescription written by the provider.

The survey study will enroll patients until December 31, 2014, or until sufficient numbers have been achieved.

Rahm Foundation will continue the study until:

* Sufficient information has accumulated to meet the scientific objectives of the Study (i.e. numeric targets or effect size)
* The feasibility of collecting sufficient information diminishes to unacceptable levels, poor enrollment, loss to follow-up and/or
* Other methods of gathering appropriate information become achievable or are deemed preferable.

Datum Research will need to have access to the prescription to see what compound was prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed a topical cream for pain, scar care, or wound OR Provider preforms urinary drug test

Exclusion Criteria:

* Subjects with legally authorized representatives
* Minors
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are given a prescription for topical compound for pain, scar care, or wound care, and agree to complete the surveys
  or
  Patients who are given a UDT and agree to complete the surveys.
  Patients will be recruited into the study if their providers prescribe a topical cream for pain, scar care or wound care or if the provider performs a UDT prior to treatment or surgery. The providers will follow their office procedure for UDT. If they perform a UDT and the patient agrees to participate in the survey study, they will have the patient complete the surveys.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain survey results from baseline at 30 days | baseline and 30 days
  Survey on pain management
Change in pain survey results from baseline at 60 days | baseline and 60 days
  Survey on pain management
Change in pain survey results from baseline at 90 days | baseline and 90 days
  Survey on pain management
Change in scar care survey results from baseline at 30 days | baseline and 30 days
  Survey on scar care
Change in scar care survey results from baseline at 60 days | baseline and 60 days
  Survey on scar care
Change in scar care survey results from baseline at 90 days | baseline and 90 days
  Survey on scar care
Change in wound care survey results from baseline at 30 days | baseline and 30 days
  Survey on wound care
Change in wound care survey results from baseline at 60 days | baseline and 60 days
  Survey on wound care
Change in wound care survey results from baseline at 90 days | baseline and 90 days
  Survey on wound care
Change in UDT survey results from baseline at 30 days | baseline and 30 days
  Survey on urinary drug testing
Change in UDT survey results from baseline at 60 days | baseline and 60 days
  Survey on urinary drug testing
Change in UDT survey results from baseline at 90 days | baseline and 90 days
  Survey on urinary drug testing

SECONDARY OUTCOMES:
Change in pain survey results from 30 days at 60 days | 30 days and 60 days
  Survey on pain management
Change in pain survey results from 30 days at 90 days | 30 days and 90 days
  Survey on pain management
Change in pain survey results from 60 days at 90 days | 60 days and 90 days
  Survey on pain management
Length of hospital stay | at baseline
  if applicable
Change in scar care survey results from 30 days at 60 days | 30 days and 60 days
  Survey on scar care
Change in scar care survey results from 30 days at 90 days | 30 days and 90 days
  Survey on scar care
Change in scar care survey results from 60 days at 90 days | 60 days and 90 days
  Survey on scar care
Change in wound care survey results from 30 days at 60 days | 30 days and 60 days
  Survey on wound care
Change in wound care survey results from 30 days at 90 days | 30 days and 90 days
  Survey on wound care
Change in UDT survey results from 60 days at 90 days | 60 days and 90 days
  Survey on urinary drug testing
Change in UDT survey results from 30 days at 60 days | 30 days and 60 days
  Survey on urinary drug testing
Change in UDT survey results from 30 days at 90 days | 30 days and 90 days
  Survey on urinary drug testing

CONTACTS AND LOCATIONS:
Locations (1):
- Blueprint Pathways, Nashville, Tennessee, United States

REFERENCES:
- See also: Blueprint Pathways — http://www.blueprintpathways.com
- See also: The Rahm Foundation — http://www.rahmfoundation.org/